CLINICAL TRIAL: NCT04332536
Title: Role and Implications of Central Fatigue Limiting Aerobic Capacity in Chronic Heart Failure: The Head vs. Heart Study
Brief Title: Limitations of Aerobic Capacity in Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Klaus K Witte, MD, Principal Investigator, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 211045
Record Dates: First submitted 2020-03-27; First posted 2020-04-02 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Chronic Heart Failure
MeSH Terms: interventions — Exercise; Codeine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chronic Heart Failure (Experimental)
  Interventions: Other: Exercise with and without Codeine
- Age-matched healthy controls (Active Comparator)
  Interventions: Other: Exercise with and without Codeine

INTERVENTIONS:
Other: Exercise with and without Codeine — This study will use our novel CPX test that incorporates instantaneous assessment of maximal isokinetic cycling power at V̇O2peak to elucidate the mechanisms that limit V̇O2peak in CHF, and compare these responses with age-matched controls.

SUMMARY:
This study will use a novel CPX test that incorporates instantaneous assessment of maximal isokinetic cycling power at V̇O2peak to elucidate the mechanisms that limit V̇O2peak in CHF, and compare these responses with age-matched controls.

DETAILED DESCRIPTION:
Chronic heart failure (CHF) is a current and growing public health concern that is expensive to treat (annual costs account for approximately 1.8% of the National Health Service budget), and associated with both poor prognosis (annual mortality ~7%) and patient quality of life. CHF is a complex, multi-faceted clinical syndrome that is characterized by profound reductions in exercise tolerance. This reduction in exercise tolerance restricts the ability to perform everyday activities such as walking, and effectively predicts declines in health-related quality of life due to symptoms of dyspnea and fatigue.

The gold-standard measure of exercise tolerance is aerobic capacity (V̇O2peak), assessed during a cycle or treadmill based exercise test. V̇O2peak is a significant predictor of cardiac-related hospitalizations and mortality risk, with every 1 ml·min-1·kg-1 reduction in V̇O2peak increasing all-cause mortality risk by ~16 %. In CHF; however, V̇O2peak is poorly related to the severity of the cardiac dysfunction. Therefore, understanding the mechanisms that limit whole-body V̇O2peak would provide novel targets for therapy, and allow for effective optimization of resource allocation to meet the needs of individual patients to ameliorate CHF symptoms, increase health-related quality of life and improve prognosis.

Treadmill and cycle ergometry cardiopulmonary exercise (CPX) tests are the gold-standard method for assessing whole-body V̇O2peak. However, the techniques currently used in clinical practice do not have the discriminatory ability to identify the fatigue mechanisms that are ultimately responsible for limiting whole-body V̇O2peak. The fatigue mechanisms limiting whole-body V̇O2peak can be defined as 'peripheral' - a reduction in the power that the exercising muscles can generate due to the accumulation of fatigue-related metabolites that impair excitation-contraction coupling; or 'central' - a reduction in skeletal muscle activation due to events within the central nervous system, the consequences of which increase the perceived effort of performing any exercise task. In essence, if peripheral fatigue limits whole-body V̇O2peak, the participant "would, but the exercising muscles can't" continue the exercise, but if central fatigue predominates, the participant "could, but won't" continue the exercise.

In young healthy participants, using a novel CPX protocol developed in our laboratory that overcomes the limitations of traditional CPX tests and allows insight into the mechanisms limiting exercise tolerance, it appears that there is an intricate coordination of peripheral and central fatigue mechanisms such that termination of the CPX test at V̇O2peak is coincident with the maximum cycling power of the legs. Thus, there is no reserve in the ability of the legs to generate cycling power at V̇O2peak, with similar findings in a healthy older population. In CHF it is often assumed that the compromised cardiac function, which reduces the ability to transport and utilize O2, accentuates the development of peripheral fatigue, with this the predominant mechanisms that limits V̇O2peak and exercise tolerance, restricting the ability to complete day-to-day activities. However, the initial cardiac event propagates a wide range of systemic effects that compromise exercise economy, skeletal muscle structure and function, and increase the ventilatory demands of any exercise task. Therefore, in CHF it is possible that these effects amplify the perceived effort of the exercise, accentuate the development of central fatigue and dissociate the normal coordination of central and peripheral fatigue mechanisms at V̇O2peak. Thus in CHF, participants may achieve V̇O2peak before peripheral fatigue has developed to the extent that this limits the ability to perform exercise, with a large reserve in the physiologic capacity of the exercising leg muscles. For the CHF patient, being able to access this reserve in the capacity of the exercising leg muscles ('power reserve') would result in clinically meaningful increases in V̇O2peak (minimally clinically important difference 1 ml·min-1·kg-1), with this expected to increase health-related quality of life.

However, central fatigue may not be the primary limitation in all CHF patients. Those with greater disease severity, longer duration of diagnosis or specific co-morbidities (e.g. type 2 diabetes) that influence the skeletal muscles may have an excessive and overriding peripheral fatigue limitation that eliminates the presence of a power reserve at V̇O2peak. For these patients, increasing V̇O2peak would be dependent on increasing physiologic capacity through interventions such as exercise rehabilitation programs.

For CHF patients in whom V̇O2peak is limited by an exaggerated central fatigue response to exercise, it is possible that acute opioid treatment may ameliorate the development of central fatigue, increasing V̇O2peak and exercise tolerance. Acute opioid treatment (dihydrocodeine) at a dose of 1 mg·kg-1 body weight reduces the perception of breathlessness, increases V̇O2peak and exercise tolerance. While it would not be expected that opioid treatment has any effect on peripheral fatigue, effects on the central nervous system may reduce the perceived effort of the exercise task and development of central fatigue. Thus opioid treatment in CHF may allow participants to 'access' a greater proportion their exercise (skeletal muscle) capacity, and evoke clinically meaningful increases in V̇O2peak and exercise tolerance. This would provide the first evidence that central fatigue can be selectively targeted in CHF to increase V̇O2peak and improve exercise tolerance. Conversely, in CHF participants in whom there is no power reserve at V̇O2peak opioid treatment would be expected to have little effect.

This study will use our novel CPX test that incorporates instantaneous assessment of maximal isokinetic cycling power at V̇O2peak to elucidate the mechanisms that limit V̇O2peak in CHF, and compare these responses with age-matched controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NYHA class I-III
* Stable CHF of at least 3 months duration
* On optimally tolerated medication for CHF
* No contraindications for cycling exercise
* Able to give informed consent

Exclusion Criteria:

* Class IV CHF
* Any contraindications to exercise
* Co-morbidities: significant COPD (FEV1<50%), severe renal disease (eGFR<20) or primary pulmonary hypertension as a co-morbidity
* Unable to give informed consent
* Current diagnosis of cancer, inflammatory or musculoskeletal disease (e.g. rheumatoid arthritis), on-going infection or sepsis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-08-25 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Maximum cycling power | One week
  Power (watts)
Power reserve at V̇O2peak | One week
  Power (watts)
V̇O2peak with opioid treatment | One week
  ml/kg/min

SECONDARY OUTCOMES:
Echocardiography | One week
  Ejection fraction
Spirometry | One week
  L/min
Electrical activity of the muscles (EMG) | One week
  Frequency
Muscle oxygenation (NIRS) | One week
  Percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-10-22): https://cdn.clinicaltrials.gov/large-docs/36/NCT04332536/SAP_000.pdf